CLINICAL TRIAL: NCT00187135
Title: Fentanyl-Propofol-EMLA or L.M.X4™ Technique for Bone Marrow Aspiration in Pediatric Patients - A Phase III Study
Brief Title: Study of Fentanyl-Propofol-EMLA of L.M.X4 Technique for Bone Marrow Aspiration
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to slow accrual.
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PFE
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Results first posted 2010-03-19 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2010-03

CONDITIONS: Bone Marrow Disease; Pain
Keywords: Pain Management; Bone Marrow Aspiration
MeSH Terms: conditions — Bone Marrow Diseases; Pain; Agnosia | interventions — Fentanyl; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Fentanyl-1mcg/kg in 3 ml of Normal Saline
  Interventions: Drug: Fentanyl; Drug: EMLA; Drug: L.M.X4; Drug: Propofol
- 2 (Active Comparator): Fentanyl - 0.5 mcg/kg in 3 ml normal saline
  Interventions: Drug: Fentanyl; Drug: EMLA; Drug: L.M.X4; Drug: Propofol
- 3 (Placebo Comparator): normal saline
  Interventions: Drug: EMLA; Drug: L.M.X4; Drug: Propofol

INTERVENTIONS:
Drug: Fentanyl — 1. Fentanyl - 1 mcg/kg in 3 ml normal saline
  2. Fentanyl - 0.5 mcg/kg in 3 ml normal saline
  Arms: 1; 2
Drug: EMLA — All patients will have EMLA or LMX4 cream applied at the anticipated site of the bone marrow aspiration to ensure topical anesthesia, and will receive a total intravenous anesthetic technique (TIVA). EMLA application has to be over at least 60 minutes and not to exceed 5 hours.
Drug: L.M.X4 — All patients will have EMLA or LMX4 cream applied at the anticipated site of the bone marrow aspiration to ensure topical anesthesia, and will receive a total intravenous anesthetic technique (TIVA). In order to optimize transdermal anesthesia LMX4 application has to be over at least 30 minutes.
Drug: Propofol — Propofol - 1 mg/kg increments every 30 seconds-1minute until loss of consciousness is indicated by lack of response to verbal command and loss of eyelid reflex.

SUMMARY:
St. Jude Children's Research Hospital is studying the best ways to prevent pain during and after procedures such as bone marrow aspiration and lumbar puncture with intrathecal (in the spinal fluid) chemotherapy. Researchers will study the effectiveness of combining anesthetics (medicines that help people sleep) and analgesics (medicines that relieve pain). Researchers believe that a combination of fentanyl (analgesic) and propofol (anesthetic), along with applying the skin-numbing-cream EMLA or L.M.X4™ on the area where the procedure is performed, will provide better pain control.

Each patient enrolled on this study will have three different anesthetic combinations for three different procedures, in order to determine which combination worked best for each child.

DETAILED DESCRIPTION:
The study focusses on the following primary aims:

* To compare 0.5 mg/kg versus 1.0 mg/kg of fentanyl to control pain in patients who have a BMT/LPIT procedure in the context of propofol anesthesia and topical anesthesia with EMLA or L•M•X 4™cream (or when necessary, lidocaine for injection).
* To compare placebo versus fentanyl (0.5 mg/kg or 1.0 mg/kg) in these same patients. The first BMT/LPIT for which patients receive any fentanyl will be used in this comparison.

The study focusses on the following secondary aims:

* To determine which dose regimen ensures best conditions to perform bone marrow aspiration (lack of motion) and maintains hemodynamic and respiratory stability as indicators of adequate levels of analgesia during bone marrow aspiration.
* To evaluate the safety and complications for each dose regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing bone marrow aspiration (unilateral), with lumbar puncture and intrathecal chemotherapy.
* Age 2 to 17 years
* ASA I-III
* Patients with acute lymphoblastic leukemia or lymphoblastic lymphoma in remission or on the day of anticipated remission procedures occurring at the end of remission induction.
* Patients must have three anticipated bone marrow aspirates and lumbar punctures with intrathecal chemotherapy remaining in their treatment

Exclusion Criteria:

* Newly diagnosed patients
* Patients with low platelet count (less than 50000)
* Patients undergoing bone marrow biopsy in addition to bone marrow aspiration
* Age less than 2 years or over 17 years
* ASA IV-V
* Patients taking opioid medication for pre-existent pain for more than 2 weeks at the time of the procedure
* Neurological impairment that would increase susceptibility to opioids (Down's syndrome)
* Clinical contraindications for general anesthesia (large mediastinal mass) or specific use of propofol, Fentanyl, EMLA, L•M•X 4™ or Lidocaine for injection

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 168 (Actual)
Dates: Start 2002-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doralina L. Anghelescu, M.D., Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 168 participants were enrolled between March, 2002 and August, 2007.
Pre-assignment Details: 168 participants were enrolled and were expected to receive 3 Bone Marrow Aspirations/Lumbar Puncture Intrathecal Chemotherapy procedures; 6 patients withdrew (eg: medical withdrawal, withdrawal of consent and other). 162 were randomized, of which 77 completed all 3 treatments.
Groups:
- Fentanyl 0.5 / Placebo / Fentanyl 1: Participants assigned to receive Fentanyl 0.5 micrograms per kilogram (mcg/kg) during their first visit, Placebo (Pl)during their second visit, and Fentanyl 1 micrograms per kilogram at the final visit.
- Fentanyl 0.5 /Fentanyl 1 / Placebo: Participants assigned to receive Fentanyl 0.5 micrograms per kilogram (mcg/kg) during their first visit, Fentanyl 1 micrograms per kilogram (mcg/kg) during their second visit, and Placebo at the final visit.
- Placebo / Fentanyl 0.5 /Fentanyl 1: Participants assigned to receive Placebo during their first visit, Fentanyl 0.5 micrograms per kilogram (mcg/kg) during their second visit, and Fentanyl 1 micrograms per kilogram (mcg/kg) at the final visit.
- Placebo /Fentanyl 1 / Fentanyl 0.5: Participants assigned to receive Placebo during their first visit, Fentanyl 1 micrograms per kilogram (mcg/kg) during their second visit, and Fentanyl 0.5 micrograms per kilogram (mcg/kg) at the final visit.
- Fentanyl 1 / Fentanyl 0.5 / Placebo: Participants assigned to receive Fentanyl 1 micrograms per kilogram (mcg/kg) during their first visit Fentanyl 0.5 micrograms per kilogram (mcg/kg) during their second visit, and Placebo at the final visit.
- Fentanyl 1 / Placebo /Fentanyl 0.5: Participants assigned to receive Fentanyl 1 micrograms per kilogram (mcg/kg) during their first visit Placebo during their second visit, and Fentanyl 0.5 micrograms per kilogram (mcg/kg) at the final visit.
Period: Visit One
Arm/Group | Fentanyl 0.5 / Placebo / Fentanyl 1 | Fentanyl 0.5 /Fentanyl 1 / Placebo | Placebo / Fentanyl 0.5 /Fentanyl 1 | Placebo /Fentanyl 1 / Fentanyl 0.5 | Fentanyl 1 / Fentanyl 0.5 / Placebo | Fentanyl 1 / Placebo /Fentanyl 0.5
Started | 30 | 28 | 25 | 26 | 25 | 28
Completed | 26 | 27 | 25 | 26 | 25 | 26
Not Completed | 4 | 1 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 3 | 1 | 0 | 0 | 0 | 1
Period: Visit Two
Arm/Group | Fentanyl 0.5 / Placebo / Fentanyl 1 | Fentanyl 0.5 /Fentanyl 1 / Placebo | Placebo / Fentanyl 0.5 /Fentanyl 1 | Placebo /Fentanyl 1 / Fentanyl 0.5 | Fentanyl 1 / Fentanyl 0.5 / Placebo | Fentanyl 1 / Placebo /Fentanyl 0.5
Started | 26 | 27 | 25 | 26 | 25 | 26
Completed | 21 | 24 | 23 | 18 | 19 | 18
Not Completed | 5 | 3 | 2 | 8 | 6 | 8
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0 | 1 | 1
Not completed — Study Discontinued | 3 | 2 | 1 | 7 | 5 | 6
Period: Visit Three
Arm/Group | Fentanyl 0.5 / Placebo / Fentanyl 1 | Fentanyl 0.5 /Fentanyl 1 / Placebo | Placebo / Fentanyl 0.5 /Fentanyl 1 | Placebo /Fentanyl 1 / Fentanyl 0.5 | Fentanyl 1 / Fentanyl 0.5 / Placebo | Fentanyl 1 / Placebo /Fentanyl 0.5
Started | 21 | 24 | 23 | 18 | 19 | 18
Completed | 14 | 17 | 14 | 9 | 11 | 12
Not Completed | 7 | 7 | 9 | 9 | 8 | 6
Not completed — Death | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 2 | 0 | 0
Not completed — Study Discontinued | 7 | 6 | 7 | 7 | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fentanyl 0.5/Placebo/Fentanyl 1 | Fentanyl 0.5/Fentanyl 1/Placebo | Placebo/Fentanyl 0.5/Fentanyl 1 | Placebo/Fentanyl 1/Fentanyl 0.5 | Fentanyl 1/Fentanyl 0.5/Placebo | Fentanyl 1/Placebo/Fentanyl 0.5 | Total
Number analyzed (Participants) | 30 | 28 | 25 | 26 | 25 | 28 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] — All 162 participants who enrolled and were randomized on the study are included in the baseline summary statistics.
  years | 6.4 (4.3) | 7.2 (4.5) | 7.6 (4.8) | 7.1 (4.1) | 7.3 (4.7) | 7.1 (4.4) | 7.1 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants] — All 162 participants who enrolled and were randomized on the study are included in the baseline summary statistics.
  Participants
    Female | 15 | 11 | 12 | 10 | 9 | 13 | 70
    Male | 15 | 17 | 13 | 16 | 16 | 15 | 92

OUTCOME MEASURES:

1. Primary Outcome: Pain(Yes/No)
Description: During the sedation recovery period, pain was measured by one of three validated pediatric scales. Scales were applied according to the developmental ability of the participant: Numerical Pain Scale, FACES pain scale, and FLACC pain scale (a score based on behaviors observed: face, legs, activity, cry, and consolability). All three scales are scored from 0 - 10 units on a scale, and are interchangeable for comparison purposes. Any score >0 was coded "pain", and score of 0 was coded "no pain", yielding one score for each participant's procedure.
Time Frame: The participant was monitored from the end of the procedure until sedation recovery, which lasted a maximum of 65 min. Discharge from the recovery area was determined by hospital standards of care.
Population: Participants in this analysis are a subset of the 162 participants randomized since not all completed 3 visits on study. If a participant completed at least Visit 2 and received each of the 2 treatments compared they are included. Treatment on each visit was randomized; therefore these numbers cannot be derived directly from the participant flow.
Measure: Number; unit: Participants
Groups:
- Fentanyl 1mcg/kg vs Placebo: Patients who completed treatment with Fentanyl 1 mcg/kg and placebo.
- Fentanyl 0.5mcg/kg vs Placebo: Patients who completed treatment with Fentanyl 0.5 mcg/kg and placebo.
Arm/Group | Fentanyl 1mcg/kg vs Placebo | Fentanyl 0.5mcg/kg vs Placebo
Number analyzed (Participants) | 71 | 79
Participants
  Pain with Fentanyl and pain with Placebo | 0 | 6
  Pain with Fentanyl and no-pain with Placebo | 7 | 8
  No-pain with Fentanyl pain with Placebo | 10 | 5
  No-pain with Fentanyl no-pain with Placebo | 54 | 60
Statistical Analysis 1: Comparison: Fentanyl 0.5mcg/kg vs Placebo; The study was designed to achieve statistical power of 80% for this comparison. Due to the early termination of the study, the sample size needed to ensure adequate statistical power for this comparison was not obtained; Test type: Superiority or Other; p = 0.5, McNemar — To adjust for multiple comparisons, p-values less than 0.0167 are considered statistically significant
Statistical Analysis 2: Comparison: Fentanyl 1mcg/kg vs Placebo; The study was designed to achieve statistical power of 80% for this comparison. The sample size needed to ensure adequate statistical power for this comparison was obtained; Test type: Superiority or Other; p = 0.5, McNemar — To adjust for multiple comparisons, p-values less than 0.0167 are considered statistically significant

2. Primary Outcome: Pain (Yes/No)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- Fentanyl 0.5mcg/kg vs Fentanyl 1mcg/kg: Patients who completed treatment with Fentanyl 0.5 mcg/kg and Fentanyl 1mcg/kg.
Arm/Group | Fentanyl 0.5mcg/kg vs Fentanyl 1mcg/kg
Number analyzed (Participants) | 74
Participants
  Pain on Fentanyl (1), Pain on Fentanyl (0.5) | 2
  Pain on Fentanyl (1) No-pain on Fentanyl (0.5) | 3
  No-Pain on Fentanyl (1), Pain on Fentanyl (0.5) | 5
  No-Pain on Fentanyl (1), No-Pain on Fentanyl (0.5) | 64
Statistical Analysis 1: Comparison: Fentanyl 0.5mcg/kg vs Fentanyl 1mcg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5, McNemar — To adjust for multiple comparisons, p-values less than 0.0167 are considered statistically significant

3. Secondary Outcome: 20% or Greater Change in Heart Rate
Description: Measurements of 20% change in Heart Rate (yes/no) taken during recovery after surgery.
Time Frame: as for outcome 1
Population: Due to study termination, not all Participants completed three planned visits. 107 of the 162 participants enrolled on study received treatment with Fentanyl 0.5 mcg/kg. 104 of the 162 participants enrolled on study received treatment with Fentanyl 1mcg/kg. 105 of the 162 participants enrolled on study received treatment with Placebo.
Measure: Number; unit: Participants
Groups:
- Fentanyl 0.5mcg/kg: Due to study termination, not all Participants completed three planned visits. Participants who completed at least one treatment with Fentanyl 0.5 mcg/kg are included in this arm. Participants were included regardless of whether they received other treatments.
- Fentanyl 1mcg/kg: Due to study termination, not all Participants completed three planned visits. Participants who completed at least one treatment with Fentanyl 1mcg/kg are included in this arm. Participants were included regardless of whether they received other treatments.
- Placebo: Due to study termination, not all Participants completed three planned visits. Participants who completed at least one treatment with Placebo are included in this arm. Participants were included regardless of whether they received other treatments.
Arm/Group | Fentanyl 0.5mcg/kg | Fentanyl 1mcg/kg | Placebo
Number analyzed (Participants) | 107 | 104 | 105
Participants
  Yes | 7 | 6 | 8
  No | 100 | 98 | 97
Statistical Analysis 1: Comparison: Fentanyl 0.5mcg/kg vs Fentanyl 1mcg/kg vs Placebo; The generalized estimation equation (GEE) approach by Liang and Zeger was used to model the effects of 20% change in heart rate (HR) on pain (Y/N) while controlling for treatment; Test type: Superiority or Other; p = 0.87, GEE Model

4. Secondary Outcome: 20% or Greater Change in Respiratory Rate
Description: Measurements of 20% change in respiratory rate(yes/no) taken during recovery after surgery.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Fentanyl 0.5mcg/kg | Fentanyl 1mcg/kg | Placebo
Number analyzed (Participants) | 107 | 104 | 105
Participants
  Yes | 21 | 20 | 24
  No | 86 | 84 | 81
Statistical Analysis 1: Comparison: Fentanyl 0.5mcg/kg vs Fentanyl 1mcg/kg vs Placebo; The generalized estimation equation (GEE) approach by Liang and Zeger was used to model the effects of 20% change in respiratory rate (RR) on pain (Y/N) while controlling for treatment; Test type: Superiority or Other; p = 0.67, GEE Model

5. Secondary Outcome: 20% or Greater Change in Blood Pressure
Description: Measurements of 20% change in blood pressure(yes/no) taken during recovery after surgery.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Number; unit: Participants
Groups:
- Placebo: Due to study termination, not all Participants completed three planned visits. Participants who completed at least one treatment with Placebo are included in this arm.
Arm/Group | Fentanyl 0.5mcg/kg | Fentanyl 1mcg/kg | Placebo
Number analyzed (Participants) | 107 | 104 | 105
Participants
  Yes | 12 | 10 | 14
  No | 95 | 94 | 91
Statistical Analysis 1: Comparison: Fentanyl 0.5mcg/kg vs Fentanyl 1mcg/kg vs Placebo; The generalized estimation equation (GEE) approach by Liang and Zeger was used to model the effects of 20% change in blood presure (BP) on pain (Y/N) while controlling for treatment; Test type: Superiority or Other; p = 0.52, GEE Model

6. Secondary Outcome: Movement
Description: Movement (yes/no) measured during recovery after surgery.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Fentanyl 0.5mcg/kg | Fentanyl 1mcg/kg | Placebo
Number analyzed (Participants) | 107 | 104 | 105
Participants
  Yes | 57 | 45 | 58
  No | 50 | 59 | 47
Statistical Analysis 1: Comparison: Fentanyl 0.5mcg/kg vs Fentanyl 1mcg/kg vs Placebo; The generalized estimation equation (GEE) approach by Liang and Zeger was used to model the effects of motion (Y/N)on pain (Y/N) while controlling for treatment; Test type: Superiority or Other; p = 0.99, GEE Model

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the time of procedure up to 7 days post procedure
Description: Four participants died during the study period.All 4 deaths were due to the primary disease or complications of the disease process.None of the deaths occurred within 7 days of that patient's procedure for which data was collected, and therefore is unrelated to the study treatment.
Groups:
- Fentanyl 1mcg/kg: Due to study termination, not all Participants completed three planned visits. Participants who completed at least one treatment with Fentanyl 1.0 mcg/kg are included in this arm. Participants were included regardless of whether they received other treatments.
Arm/Group | Fentanyl 0.5mcg/kg | Fentanyl 1mcg/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/107 | 0/104 | 0/105
Other Adverse Events (participants affected / at risk) | 0/107 | 0/104 | 0/105

LIMITATIONS AND CAVEATS:
All 162 participants were expected to receive three treatments. Not all participants received all three treatments. Therefore, analysis required the identification of subsets of treated participants. The trial terminated early due to slow accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes